CLINICAL TRIAL: NCT00001656
Title: Childhood Onset Psychotic Disorders: Characterization and Treatment With Atypical Neuroleptics
Brief Title: Comparison of Clozapine vs Olanzapine in Childhood-Onset Psychotic Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Judith L. Rapoport, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 970126; 97-M-0126
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-03

CONDITIONS: Childhood Schizophrenia; Psychotic Disorder; Schizophrenia
Keywords: Clozapine; Olanzapine; Drug Response; Safety; Childhood Onset Schizophrenia; Schizoaffective Disorder; Multidimensionally Impaired Syndrome; Phenomenology; Biochemical Correlates; Brain Imaging; Schizophrenia; Childhood Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia, Childhood; Psychotic Disorders; Schizophrenia | interventions — Olanzapine; Clozapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine
- Clozapine (Active Comparator)
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Olanzapine — tablet; 5-20mg/day; 8 weeks
  Other Names: "Zyprexa"
  Arms: Olanzapine
Drug: Clozapine — tablet; 12.5-900mg/day; 8 weeks
  Other Names: "Clozaril"
  Arms: Clozapine

SUMMARY:
The purpose of this study is to compare the effectiveness and side effects of the drugs clozapine and olanzapine in children and adolescents with schizophrenia and psychoses.

Childhood psychosis is a serious disorder that may have devastating consequences. Effective treatments for the condition are under continual investigation. This study will examine the causes of and offer treatment for childhood psychosis.

Participants in this study will undergo psychological tests, blood and urine tests, electroencephalogram (EEG), electrocardiogram (EKG), and magnetic resonance imaging (MRI) scans of the brain for the first 1 to 2 weeks of the study while taking their regular medications. Participants will then be tapered off their medications over 1 to 3 weeks and will continue to stay off medications for an additional 2 days to 3 weeks. During this time, participants will undergo psychiatric, neurological, and cardiac examinations as well as blood tests. After this period without medications, participants will be randomly assigned to receive either clozapine or olanzapine for 8 weeks. An EEG will be performed prior to treatment and after 6 weeks of study medication. Participants who respond well to the study drugs may continue to receive them through their own physician. Participants who do not respond to either clozapine or olanzapine or cannot tolerate their side effects will be treated individually with other drugs until optimum treatment is identified. Regular telephone updates and in person visits to NIH for repeat testing and MRIs will be conducted.

DETAILED DESCRIPTION:
The purpose of this protocol is to compare efficacy of clozapine and olanzapine in children and adolescents with schizophrenia and psychoses, as well as to learn about side effects of these medication in pediatric population. The underlying hypothesis is that clozapine has superior efficacy over olanzapine.

Children and adolescents, ages 7 to 18 years, meeting DSM-IV criteria for schizophrenia, schizoaffective disorder and psychotic disorder not otherwise specified, with onset of psychosis before their 13th birthday, who have not responded to at least two prior trials with typical or a typical neuroleptics, will be eligible to participate in a double-blind, parallel group, trial of olanzapine-clozapine.

This study will be done in conjunction with the Screening protocol, which will include characterization by clinical phenomenology, eye tracking, MRI brain imaging, plasma biochemistry, and chromosomal analysis.

This study will consist of the following phases 1) Tapering of psychotropic medications (1-4 weeks, depending upon type and dosage). 2) Observation for up to 2 weeks drug free, in order to establish a baseline prior to starting medication trial. 3) An 8 week double-blind trial of either clozapine or olanzapine. Efficacy and tolerability of clozapine and olanzapine will be compared using specified criteria. 4) If desired improvement not achieved or trial is interrupted, an 8 week open trial of the second medication and 5) Discharge following medication optimization for up to 4 weeks, or as clinically appropriate. This protocol also includes a follow-up every 2 to 3 years for a period of 10 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males and females, age 7 to 18 years

Onset of psychotic symptoms before 13th birthday and a DSM-IV diagnosis of either schizophrenia, schizoaffective disorder, MDI syndrome, or psychosis NOS (not otherwise specified).

Current significant impairment due to the illness (current psychotic symptoms, decline of functioning academically and socially, significant discomfort due to psychotic symptoms).

Failure of two prior trials with antipsychotic medications (either typical or atypical) used at adequate doses (greater than or equal to 100 mg/day in chlorpromazine equivalents) and for adequate duration (at least 4 weeks, unless terminated due to intolerable side effects). Failure is defined as either insufficient response with persistence of symptoms significantly impairing child's functioning, according to child's and parental reports and medical and school records, or intolerable side effects to drugs other than clozapine and olanzapine.

Subjects may be included if their previous trial(s) of olanzapine failed to reach the dose of 20. mg/day or a duration of fewer than four weeks.

Subjects may be included if their previous trial(s) of clozapine failed to reach the dose of 200. mg/day or a duration of fewer than six weeks.

Comorbid psychiatric disorders in the past 12 months are permitted as long as not clinically significant.

EXCLUSION CRITERIA:

Prepsychotic full-scale IQ less than 70.

Unstable major neurological or medical conditions.

Current pregnancy or plan to become pregnant during the first three months (the duration of the study) in woman of childbearing age; breast-feeding in woman with infants.

DSM-IV substance abuse or dependence in the past 6 months.

True non-responders to either olanzapine or clozapine. True non-response is defined as: a) intolerance to either of the medications preventing an adequate trial, or b) only minimal (less than 20%) benefit with the adequate trial of either of the medications. Adequate trial constitutes at least 8 weeks of the medication with the dose of 20 mg on olanzapine or 200 mg of clozapine.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 1997-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Rapoport, M.D., Principal Investigator — Child Psychiatry Branch, NIMH, NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gordon CT, Frazier JA, McKenna K, Giedd J, Zametkin A, Zahn T, Hommer D, Hong W, Kaysen D, Albus KE, et al. Childhood-onset schizophrenia: an NIMH study in progress. Schizophr Bull. 1994;20(4):697-712. doi: 10.1093/schbul/20.4.697. PMID 7701277
- [Background] Nicolson R, Rapoport JL. Childhood-onset schizophrenia: rare but worth studying. Biol Psychiatry. 1999 Nov 15;46(10):1418-28. doi: 10.1016/s0006-3223(99)00231-0. PMID 10578456
- [Result] Shaw P, Sporn A, Gogtay N, Overman GP, Greenstein D, Gochman P, Tossell JW, Lenane M, Rapoport JL. Childhood-onset schizophrenia: A double-blind, randomized clozapine-olanzapine comparison. Arch Gen Psychiatry. 2006 Jul;63(7):721-30. doi: 10.1001/archpsyc.63.7.721. PMID 16818861
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_1997-M-0126.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine Group; Clozapine Group: All medications were given by mouth, in identical tablet form. Day 1, patient was given 5mg olanzapine or 12.5mg clozapine. Clozapine dose was then increased every other day, the first increase by 12.5mg (to a total dose of 25mg/day) and then in steps of 25mg. When the clozapine dose reached 150mg/day, the olanzapine dose was increased to 10mg/day. When the clozapine dose reached 300mg/day, the olanzapine dose was increased to 15mg/day. Further increases were guided by clinical judgment to a maximum of 20mg/day of olanzapine and 900mg/day of clozapine.
Period: Overall Study
Arm/Group | Olanzapine Group | Clozapine Group
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine Group | Clozapine Group | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 12 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.8 (2.4) | 11.7 (2.3) | 12.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 7 | 8 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in the Scale for the Assessment of Negative Symptoms
Description: Measures change in affective flattening or blunting, alogia, avolition/apathy, anhedonia/asociality, attention; minimum score = 0; maximum score = 125; lower values are considered a better outcome
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | -14 [-20 to -7] | -25 [-34 to -15]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Analysis of covariance with baseline score as covariate; Test type: Superiority or Other; p = .04, ANCOVA; Covariate is baseline score

2. Primary Outcome: Change in the Clinical Global Impression Severity of Symptoms Scale
Description: Measures change in the severity of symptoms; Minimum score = 1; maximum score = 7; lower score is considered a better outcome.
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | -0.6 [-1.3 to 0.1] | -1.6 [-2.3 to -0.8]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Analysis of covariance with baseline score as covariate; Test type: Superiority or Other; p = 0.21, ANCOVA; Covariate is baseline score

3. Primary Outcome: Change in the Brief Psychiatric Rating Scale-24
Description: A 24-item scale measuring change in interpersonal behaviors, mood, psychosis, anxiety, speech, sleep, orientation and physical activity. Lowest score = 24; highest score = 168; lower score is considered a better outcome.
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | -13 [-21 to -6] | -19 [-26 to -12]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Analysis of covariance with baseline score as covariate; Test type: Superiority or Other; p = 0.35, ANCOVA

4. Primary Outcome: Change in the Scale for the Assessment of Positive Symptoms
Description: Measures change in hallucinations, delusions, bizarre behavior, and thought organization. Minimum score = 0; maximum score = 170; lower score is considered a better outcome.
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | -7 [-18 to 5] | -21 [-33 to -9]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Analysis of covariance with baseline score as covariate; Test type: Superiority or Other; p = 0.19, ANCOVA; Covariate is baseline score

5. Primary Outcome: Change in the Bunney-Hamburg Rating Scale for Psychosis
Description: Measures change in psychosis severity; Minimum score = 0; maximum score = 7; lower score is considered a better outcome.
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | -3.1 [-5.0 to -1.2] | -4 [-5.3 to -2.7]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Analysis of covariance with baseline score as covariate; Test type: Superiority or Other; p = 0.59, ANCOVA; Covariate is baseline score

6. Primary Outcome: Change in Bunney-Hamburg Rating Scale for Depression
Description: Measures change in severity of depression; Minimum score = 0; maximum score = 7; lower score is considered a better outcome.
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | 0.4 [-0.6 to 1.4] | 0.2 [-0.5 to 0.8]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Analysis of covariance with baseline score as covariate; Test type: Superiority or Other; p = 0.72, ANCOVA

7. Primary Outcome: Change in Bunney-Hamburg Rating Scale for Mania
Description: Measures change in the severity of mania; Minimum score = 0; maximum score = 7; lower score is considered a better outcome.
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | -0.4 [-2.3 to 1.5] | -0.8 [-1.7 to 0.1]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Analysis of covariance with baseline score as covariate; Test type: Superiority or Other; p = 0.27, ANCOVA; Covariate is baseline score

8. Primary Outcome: Change in the Bunney-Hamburg Rating Scale for Anxiety
Description: Measures change in the severity of anxiety; Minimum score = 0; maximum score = 7; lower score is considered a better outcome.
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
Scores on a scale | -0.5 [-1.6 to 0.5] | 0.6 [-2.3 to 1.1]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Test type: Superiority or Other; p = 0.11, ANCOVA; Covariate is baseline score

9. Other Pre Specified Outcome: Change in Weight
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
kilograms | 3.6 (4.0) | 3.8 (6.0)
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Test type: Superiority or Other; p = 0.96, t-test, 2 sided

10. Other Pre Specified Outcome: Change in Body Mass Index (BMI)
Description: BMI is calculated by the following formula: weight (in kilograms) divided by the square of the height (in meters)
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
kg/m² | 1.4 (1.6) | 1.6 (2.5)
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Test type: Superiority or Other; p = 0.76, t-test, 2 sided

11. Other Pre Specified Outcome: Change in Extrapyramidal Movements as Measured by the Abnormal Involuntary Movements Scale (AIMS)
Description: minimum score = 10; maximum score = 50; lower score is considered a more favorable outcome
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
scores on a scale | 0 [-9 to 4] | 0 [-4 to 8]

12. Other Pre Specified Outcome: Change in Extrapyramidal Movements as Measured by the Simpson Angus Scale Score
Description: minimum score = 10; maximum score = 90; lower score considered a more favorable outcome
Time Frame: 8 week double-blind study period; baseline and 8 weeks
Measure: Median (95% Confidence Interval); unit: scores on a scale
Arm/Group | Olanzapine Group | Clozapine Group
Number analyzed (Participants) | 13 | 12
scores on a scale | 0 [-2 to 1] | 0 [-3 to 1]
Statistical Analysis 1: Comparison: Olanzapine Group vs Clozapine Group; Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 8 week-double-blind study period
Description: All adverse side effects are reported.
Arm/Group | Olanzapine Group | Clozapine Group
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine Group (N=13) | Clozapine Group (N=12)
Abnormal white blood count (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — Total white blood count > 2000; absolute neutrophil count between 1000 and 1500
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olanzapine Group (N=13) | Clozapine Group (N=12)
Enuresis (Renal and urinary disorders) | 1 (1) | 5 (5)
Increased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hypersalivation (Gastrointestinal disorders) | 4 (4) | 8 (8)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Difficulty concentrating (Nervous system disorders) | 1 (1) | 4 (4)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2)
Insomnia (Nervous system disorders) | 1 (1) | 3 (3)
Hypertension (Cardiac disorders) | 1/11 (1) | 7/11 (7)
tachycardia >100 beats/min (supine) (Cardiac disorders) | 2/12 (2) | 7/10 (7)
Tachycardia >120 beats/min (supine) (Cardiac disorders) | 0/12 (0) | 1/10 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes